CLINICAL TRIAL: NCT00667355
Title: A Multi-Center, Open-Label Efficacy, Safety, and Pharmacokinetic Study of Adalimumab in Japanese Subjects With Active Ankylosing Spondylitis
Brief Title: A Study of Adalimumab in Japanese Subjects With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-239
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2010-08-11 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab (Experimental): Adalimumab 40 mg or 80 mg subcutaneously (SC) administered every other week (eow) until approval of adalimumab for Ankylosing Spondylitis (AS) in Japan. All subjects received 40 mg of adalimumab SC eow at Baseline. The subjects who completed 16 weeks of therapy and who failed to achieve Assessments in Ankylosing Spondylitis 20 (ASAS 20) response on or after Week 16, could increase the dose of adalimumab to 80 mg eow. When the dose was increased, the higher dose was to be continued during the rest of the study.
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — 40 mg or 80 mg every other week, subcutaneous
  Other Names: ABT-D2E7; Humira

SUMMARY:
To evaluate efficacy, safety and pharmacokinetics of adalimumab in Japanese subjects with active ankylosing spondylitis

DETAILED DESCRIPTION:
It is reported that the prevalence of Ankylosing Spondylitis (AS) in Japanese patients is extremely lower than that of Caucasians; therefore, a controlled, double-blind study with similar sample size in Western studies for active AS in Japan was not able to be conducted. As a result, this study was conducted with an open-label design to investigate efficacy, safety and pharmacokinetics of adalimumab in Japanese subjects with active AS. The inclusion criteria and primary endpoint measurement (Achieving Assessment in Ankylosing Spondylitis 20 at Week 12) were designed the same as the Western studies for active AS in consideration with the confirmation of Western data. Treatment with adalimumab was to be continued until the approval of adalimumab for AS in Japanese subjects with active AS.

ELIGIBILITY:
Inclusion Criteria:

* Subject who meets the definition of Ankylosing Spondylitis based on the Modified New York Criteria, has a diagnosis of active Ankylosing Spondylitis and has had an inadequate response to or intolerance to one or more nonsteroidal anti-inflammatory drugs

Exclusion Criteria:

* History of cancer, lymphoma, leukemia or lymphoproliferative disease, active TB, HIV
* Previously received anti-TNF therapy
* Spinal surgery or joint surgery involving joints to be assessed within 2 months prior to the Screening

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hideyuki Hashiba, BS, Study Director — Abbott
Locations (19):
- Japan (19):
  - Site Reference # / Investigator 46791, Aichi
  - Site Reference # / Investigator 46789, Fukui
  - Site Reference # / Investigator 46798, Fukuoka
  - Site Reference # / Investigator 46799, Fukuoka
  - Site Reference # / Investigator 46796, Hiroshima
  - Site Reference # / Investigator 46782, Hokkaido
  - Site Reference # / Investigator 7297, Hokkaido
  - Site Reference # / Investigator 46795, Hyōgo
  - Site Reference # / Investigator 46797, Kagawa
  - Site Reference # / Investigator 46787, Kanagawa
  - Site Reference # / Investigator 46790, Nagano
  - Site Reference # / Investigator 46793, Osaka
  - Site Reference # / Investigator 46794, Osaka
  - Site Reference # / Investigator 46783, Saitama
  - Site Reference # / Investigator 46784, Saitama
  - Site Reference # / Investigator 46792, Shiga
  - Site Reference # / Investigator 46785, Tokyo
  - Site Reference # / Investigator 46786, Tokyo
  - Site Reference # / Investigator 46788, Toyama

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Adalimumab 40 mg or 80 mg subcutaneously administered every other week until approval of adalimumab for Ankylosing Spondylitis (AS) in Japan.
Period: Overall Study
Arm/Group | Adalimumab
Started | 41
Completed | 30
Not Completed | 11
Not completed — Adverse Event | 5
Not completed — Lost to Follow-up | 1
Not completed — Other reason was not specified | 5

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
Age, Customized [Number; unit: subjects]
  <40 years | 25
  Between 40 and 65 years | 16
  >65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.2 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 32
Region of Enrollment [Number; unit: subjects]
  Japan | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Assessment in Ankylosing Spondylitis 20 (ASAS 20) at Week 12
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) subjects. ASAS has 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 20 = at least 20% improvement (vs. baseline) and an absolute improvement ≥ 10 units on a 0 - 100 scale (0 = no disease activity; 100 = high disease activity) for ≥ 3 domains, and no worsening (defined as a worsening of ≥ 20% and a net worsening of ≥ 10 units) in the remaining domain.
Time Frame: Week 12
Population: For all non-responder imputation (NRI) analyses, subjects with a missing value at a visit were imputed as a non-responder for that visit. Observed cases is based on a total of 40 subjects analyzed (vs. 41 subjects for the study and all other analysis sets) due to 1 subject who discontinued prior to Week 12.
Measure: Number; unit: Subjects
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
Subjects
  Non-responder imputation (NRI), N = 41 | 30
  Last Observation Carried Forward (LOCF), N = 41 | 30
  Observed Cases, N = 40 | 30

2. Secondary Outcome: Number of Subjects Achieving ASAS 20
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) subjects. ASAS has 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 20 = 20% improvement (vs. baseline) and an absolute improvement ≥ 10 units on a 0-100 scale (0 = no disease activity; 100 = high disease activity) for ≥ 3 domains, and no worsening (defined as a worsening of ≥ 20% and a net worsening of ≥ 10 units) in the remaining domain.
Time Frame: Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on non-responder imputation (NRI), for which subjects with a missing value at a visit were imputed as a non-responder for that visit.
Measure: Number; unit: Subjects
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
Subjects
  Week 12 | 30
  Week 24 | 30
  Week 48 | 32
  Week 72 | 32
  Week 96 | 27
  Week 120 | 21
  Final Visit | 32

3. Secondary Outcome: Number of Subjects Achieving ASAS 50
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) subjects. ASAS has 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 50 = at least 50% improvement (vs. baseline) and an absolute improvement ≥ 20 units on a 0-100 scale (0 = no disease activity; 100 = high disease activity) for ≥ 3 domains, and no worsening (defined as a worsening of ≥ 20% and a net worsening of ≥ 10 units) in the remaining domain.
Time Frame: Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on NRI, for which subjects with a missing value at a visit were imputed as a non-responder for that visit.
Measure: Number; unit: Subjects
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
Subjects
  Week 12 | 23
  Week 24 | 26
  Week 48 | 26
  Week 72 | 25
  Week 96 | 19
  Week 120 | 17
  Final Visit | 27

4. Secondary Outcome: Number of Subjects Achieving ASAS 70
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) subjects. ASAS has 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 70 = at least 70% improvement (vs. baseline) and an absolute improvement ≥ 30 units on a 0-100 scale (0 = no disease activity; 100 = high disease activity) for ≥ 3 domains, and no worsening (defined as a worsening of ≥ 20% and a net worsening of ≥ 10 units) in the remaining domain.
Time Frame: Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
Subjects
  Week 12 | 13
  Week 24 | 16
  Week 48 | 18
  Week 72 | 17
  Week 96 | 15
  Week 120 | 13
  Final Visit | 19

5. Secondary Outcome: Number of Subjects Achieving Bath Ankylosing Spondylitis Disease Activity Index 50 (BASDAI 50)
Description: BASDAI is a validated self assessment tool used to determine disease activity in subjects with Ankylosing Spondylitis (AS). Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) subjects answered 6 questions measuring discomfort, pain, fatigue, and morning stiffness. BASDAI 50 = at least 50% improvement (vs. baseline) in BASDAI.
Time Frame: Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
Subjects
  Week 12 | 27
  Week 24 | 26
  Week 48 | 25
  Week 72 | 28
  Week 96 | 22
  Week 120 | 18
  Final Visit | 29

6. Secondary Outcome: Mean Change From Baseline in Patient's Global Assessment of Disease Activity
Description: Subject's assessment of disease activity using a Visual Analog Scale (VAS) of 0 - 100 mm (0 = none and 100 = severe).
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on LOCF.
Measure: Mean (95% Confidence Interval); unit: mm on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
mm on scale
  Week 12 | -34.6 [-42.80 to -26.33]
  Week 24 | -37.3 [-45.99 to -28.69]
  Week 48 | -39.5 [-47.52 to -31.51]
  Week 72 | -39.7 [-48.14 to -31.32]
  Week 96 | -37.1 [-45.96 to -28.34]
  Week 120 | -40.1 [-48.61 to -31.53]
  Final Visit | -40.6 [-48.81 to -32.32]

7. Secondary Outcome: Mean Change From Baseline in Total Back Pain
Description: Subject assessed his/her back pain by using a Visual Analog Scale (VAS) of 0 - 100 mm (0 = no pain and 100 = most severe pain).
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on LOCF.
Measure: Mean (95% Confidence Interval); unit: mm on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
mm on scale
  Week 12 | -35.6 [-43.68 to -27.59]
  Week 24 | -37.0 [-45.05 to -28.85]
  Week 48 | -38.6 [-46.68 to -30.53]
  Week 72 | -39.3 [-47.53 to -31.01]
  Week 96 | -36.4 [-44.33 to -28.40]
  Week 120 | -39.2 [-46.98 to -31.36]
  Final Visit | -40.2 [-47.80 to -32.64]

8. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: BASFI is a validated self assessment tool that determines the degree of functional limitation in AS subjects. Utilizing a VAS of 0-100 mm (0=easy, 100=impossible), subjects answered 10 questions assessing their ability in completing normal daily activities or physically demanding activities. The BASFI score is a mean score of the 10 questions.
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on last observation carried forward (LOCF).
Measure: Mean (95% Confidence Interval); unit: mm on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
mm on scale
  Week 12 | -19.4 [-24.49 to -14.34]
  Week 24 | -20.5 [-25.84 to -15.08]
  Week 48 | -21.9 [-28.39 to -15.51]
  Week 72 | -22.2 [-29.44 to -14.89]
  Week 96 | -22.1 [-28.72 to -15.54]
  Week 120 | -21.8 [-28.07 to -15.51]
  Final Visit | -21.6 [-27.65 to -15.49]

9. Secondary Outcome: Mean Change From Baseline in C-Reactive Protein (CRP)
Description: CRP is a marker of inflammation and measured in mg/dL. A higher level is consistent with inflammation.
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on LOCF.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
mg/dL
  Week 12 | -1.2 [-1.60 to -0.83]
  Week 24 | -1.3 [-1.76 to -0.89]
  Week 48 | -1.4 [-1.78 to -0.95]
  Week 72 | -1.3 [-1.74 to -0.83]
  Week 96 | -1.4 [-1.84 to -0.94]
  Week 120 | -1.3 [-1.76 to -0.76]
  Final Visit | -1.2 [-1.67 to -0.64]

10. Secondary Outcome: Number of Subjects Achieving Assessment in Ankylosing Spondylitis (ASAS) 5/6.
Description: ASAS 5/6 consists of 6 domains: the 4 used in ASAS 20 (patient global assessment of disease activity, pain, function, inflammation) plus spinal mobility and an acute phase reactant, C Reactive Protein (CRP). Achieving ASAS 5/6 requires a 20% improvement compared to baseline in ≥ 5 domains (each domain measured on a 0 - 100 scale [0 = no disease activity; 100 = high disease activity]).
Time Frame: Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
Subjects
  Week 12 | 28
  Week 24 | 29
  Week 48 | 31
  Week 72 | 28
  Week 96 | 25
  Week 120 | 20
  Final Visit | 29

11. Secondary Outcome: Number of Subjects Achieving Assessment in Ankylosing Spondylitis 40 (ASAS 40)
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) subjects. ASAS = 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 40 = at least 40% improvement (vs. baseline) and an absolute improvement ≥ 20 units on a 0-100 scale (0 = no disease activity; 100 = high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
Subjects
  Week 12 | 26
  Week 24 | 26
  Week 48 | 27
  Week 72 | 28
  Week 96 | 24
  Week 120 | 18
  Final Visit | 26

12. Secondary Outcome: Number of Subjects Achieving Assessment in Ankylosing Spondylitis Partial Remission
Description: Partial remission is defined as a score of less than 20 units (on a scale of 0-100; 0=no disease activity and 100=high disease activity) in each of the 4 Assessments in Ankylosing Spondylitis (ASAS) domains: patient global assessment of disease activity, pain, function, and inflammation.
Time Frame: Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
Subjects
  Week 12 | 15
  Week 24 | 16
  Week 48 | 17
  Week 72 | 20
  Week 96 | 15
  Week 120 | 13
  Final Visit | 19

13. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: tragus to wall distance, lumbar flexion, cervical rotation, lumbar side flexion, and intermalleolar distance. Each measure was scored 0-2 (0=normal mobility/mild disease involvement, 1=moderate disease involvement, 2=severe disease involvement) to give a final total score ranging from 0 to 10. The higher the BASMI score, the more severe was the subject's limitation of movement due to their AS.
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
units on scale
  Week 12 | -0.4 [-0.79 to -0.02]
  Week 24 | -0.5 [-0.90 to -0.17]
  Week 48 | -0.6 [-1.07 to -0.23]
  Week 72 | -0.5 [-0.95 to -0.06]
  Week 96 | -0.6 [-1.03 to -0.13]
  Week 120 | -0.7 [-1.09 to -0.22]
  Final Visit | -0.6 [-1.00 to -0.21]

14. Secondary Outcome: Mean Change From Baseline in Chest Expansion
Description: Chest expansion is the difference in centimeters between full expiration and full inspiration, measured at the 4th inter-costal space. An increase in chest expansion represents improvement.
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on LOCF.
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
cm
  Week 12 | 0.7 [0.30 to 1.03]
  Week 24 | 0.4 [0.16 to 0.66]
  Week 48 | 0.8 [0.40 to 1.17]
  Week 72 | 1.0 [0.56 to 1.46]
  Week 96 | 0.6 [0.19 to 1.11]
  Week 120 | 1.1 [0.55 to 1.72]
  Final Visit | 1.2 [0.54 to 1.80]

15. Secondary Outcome: Mean Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
Description: Assessment of enthesitis was performed in the following 7 domains: 1) 1st costochondral joint left and right, 2) 7th costochondral joint left and right, 3) posterior superior iliac spine left and right, 4) anterior superior iliac spine left and right, 5) iliac crest left and right, 6) 5th lumbar spinous process and 7) proximal insertion of Achilles tendon left and right. Each domain was graded for the presence (1) and absence (0) of tenderness yielding total MASES ranging from 0 (no tenderness) to 13 (worst possible score; severe tenderness).
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on LOCF.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
units on a scale
  Week 12 | -1.0 [-1.71 to -0.39]
  Week 24 | -1.1 [-1.76 to -0.53]
  Week 48 | -1.3 [-1.90 to -0.74]
  Week 72 | -1.1 [-1.72 to -0.48]
  Week 96 | -1.4 [-1.98 to -0.85]
  Week 120 | -1.4 [-1.96 to -0.77]
  Final Visit | -1.4 [-1.96 to -0.77]

16. Secondary Outcome: Mean Change From Baseline in Nocturnal Pain
Description: Nocturnal pain assessed by subjects using a Visual Analog Scale (VAS) of 0 - 100 mm (0 = no pain and 100 = worst possible pain).
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on LOCF.
Measure: Mean (95% Confidence Interval); unit: mm on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
mm on scale
  Week 12 | -30.0 [-39.71 to -20.29]
  Week 24 | -31.7 [-41.92 to -21.54]
  Week 48 | -35.8 [-45.04 to -26.61]
  Week 72 | -34.6 [-43.45 to -25.77]
  Week 96 | -33.4 [-43.14 to -23.69]
  Week 120 | -35.0 [-44.10 to -25.85]
  Final Visit | -35.3 [-44.52 to -26.07]

17. Secondary Outcome: Mean Change From Baseline in Swollen Joint Count for 44 Joints (SJC 44)
Description: The number of swollen joints among 22 anatomical joints for both the right and left side of the body were assessed by a joint evaluator where the presence of a swollen joint was scored as 1 and absence as 0. The total SJC was derived by the sum of the scores for a range of SJC from 0 (best possible score; no swollen joints) to 44 (worse possible score; all joints swollen).
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on LOCF.
Measure: Mean (95% Confidence Interval); unit: SJC
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
SJC
  Week 12 | -1.1 [-1.91 to -0.38]
  Week 24 | -1.1 [-1.81 to -0.34]
  Week 48 | -1.1 [-1.97 to -0.32]
  Week 72 | -1.3 [-2.17 to -0.37]
  Week 96 | -1.2 [-1.99 to -0.44]
  Week 120 | -1.2 [-2.01 to -0.43]
  Final Visit | -1.2 [-1.94 to -0.40]

18. Secondary Outcome: Mean Change From Baseline in Tender Joint Count for 46 Joints (TJC 46)
Description: The number of tender or painful joints among 23 anatomical joints for both the right and left side of the body were assessed by a joint evaluator where the presence of a tender or painful joint was scored as 1 and absence as 0. The total TJC was derived by the sum of the scores for a range of TJC from 0 (best possible score; no tender or painful joints) to 46 (worst possible score; all joints tender or painful).
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on LOCF.
Measure: Mean (95% Confidence Interval); unit: TJC
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
TJC
  Week 12 | -1.5 [-3.86 to 0.94]
  Week 24 | -1.4 [-3.66 to 0.87]
  Week 48 | -1.3 [-3.60 to 0.96]
  Week 72 | -1.6 [-4.00 to 0.88]
  Week 96 | -1.6 [-3.63 to 0.46]
  Week 120 | -1.6 [-3.69 to 0.56]
  Final Visit | -1.6 [-3.69 to 0.56]

19. Secondary Outcome: Mean Change From Baseline in 36-Item Short Form (SF-36) Questionnaire
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These are summarized in a physical component summary (PCS) and mental component summary (MCS) score. The score for a section is an average of the individual question scores, which are scaled 0-100 (0=lowest level of functioning; 100=highest level of functioning).
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, and Final Visit
Population: Analysis is based on LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 41
units on scale
  PCS Week 12 | 9.6 [6.81 to 12.40]
  PCS Week 24 | 10.6 [7.51 to 13.67]
  PCS Week 48 | 11.4 [8.69 to 14.06]
  PCS Week 72 | 11.3 [8.29 to 14.30]
  PCS Week 96 | 12.3 [9.25 to 15.37]
  PCS Week 120 | 12.1 [9.07 to 15.19]
  PCS Final Visit | 12.6 [9.75 to 15.53]
  MCS Week 12 | 7.0 [3.07 to 10.87]
  MCS Week 24 | 7.0 [3.62 to 10.34]
  MCS Week 48 | 6.1 [2.52 to 9.59]
  MCS Week 72 | 6.7 [2.94 to 10.53]
  MCS Week 96 | 5.8 [2.55 to 9.09]
  MCS Week 120 | 6.1 [2.63 to 9.59]
  MCS Final Visit | 5.9 [2.44 to 9.42]

ADVERSE EVENTS:
Time Frame: All adverse events reported from the time of first study drug administration until 70 days following discontinuation of study drug administration were collected.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 6/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=41)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Intervertebral discitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cataract (Eye disorders) | 2
Periodontitis (Gastrointestinal disorders) | 1
Septic shock (Infections and infestations) | 1
Adenomyosis (Reproductive system and breast disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=41)
Cataract (Eye disorders) | 4
Conjunctivitis allergic (Eye disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 3
Injection site erythema (General disorders) | 6
Hepatic function abnormal (Hepatobiliary disorders) | 9
Hepatic steatosis (Hepatobiliary disorders) | 3
Nasopharyngitis (Infections and infestations) | 22
Upper respiratory tract infection (Infections and infestations) | 8
Pharyngitis (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 3
Weight increased (Investigations) | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 3
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 8
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 7
Contusion (Injury, poisoning and procedural complications) | 6
Influenza (Infections and infestations) | 4
Nausea (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
C-reactive protein increased (Investigations) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 3
Malaise (General disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Rhinitis (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements vary; the Medical Institution shall not disclose any material/information disclosed by Abbott Japan in connection with the Clinical Research or information obtained by conducting the Clinical Research to third parties without Abbott Japan's prior written approval. When Medical Institution intends to publish information obtained by conducting Clinical Research, Institution shall obtain Abbott Japan's prior written approval.